CLINICAL TRIAL: NCT02069808
Title: Efficacy of Recombinant FSH/GnRH Antagonist Protocol With and Without LH Adjunct and GnRH Agonist Trigger for Egg Bank Donation
Brief Title: Efficacy of Recombinant FSH/GnRH Antagonist Protocol With and Without LH Adjunct for Egg Bank Donation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michigan Reproductive Medicine (Other)
Responsible Party: Principal Investigator, Michael S. Mersol-Barg, MD, Principle Investigator, Michigan Reproductive Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRM2014-1
Record Dates: First submitted 2014-02-19; First posted 2014-02-24 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Egg Donation
MeSH Terms: interventions — follitropin beta; Glycoprotein Hormones, alpha Subunit; ganirelix; Menotropins; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group B: Follistim and Menopur (Experimental): Group B: N=25 subjects
  1. Cycle day 2 start Follistim 200 U/day up to 11 days duration.
  2. Cycle day 2 start Menopur (menotropins) 75 U/day up to 11 days duration.
  3. Add GnRH antagonist Ganirelix 250 µg/day starting 5 days before GnRH agonist trigger.
  4. GnRH agonist Leuprolide Acetate (Lupron) 1 mg subcutaneous injection 36 hours prior to egg collection.
  5. Transvaginal ultrasound guided needle aspiration of oocytes 36 hours after Lupron trigger.
  Interventions: Drug: Follistim; Drug: Ganirelix; Drug: Menotropins; Drug: Leuprolide; Procedure: Transvaginal ultrasound guided needle aspiration of oocytes
- Group A: Follistim only (Active Comparator): Group A: N=25 subjects
  1. Cycle day 2 start Follistim 250 U/day up to 11 days duration.
  2. Add GnRH antagonist Ganirelix 250 µg/day starting 5 days before GnRH agonist trigger.
  3. GnRH agonist Leuprolide Acetate (Lupron) 1 mg subcutaneous injection 36 hours prior to egg collection.
  4. Transvaginal ultrasound guided needle aspiration of oocytes 36 hours after Lupron trigger.
  Interventions: Drug: Follistim; Drug: Ganirelix; Drug: Leuprolide; Procedure: Transvaginal ultrasound guided needle aspiration of oocytes

INTERVENTIONS:
Drug: Follistim — Follicle stimulating hormone promotes recruitment of follicles for ovulation.
  Other Names: Follistim AQ
Drug: Ganirelix — GnRH antagonist preventing a problematic risk of premature LH surge during ovulation induction therapy.
  Other Names: Ganirelix Acetate
Drug: Menotropins — Combination of follicle stimulating hormone and Luteinizing hormone activity promotes recruitment of follicles for ovulation. Absence or presence of this medication is the difference being tested between the two arms of the study.
  Other Names: Menopur
  Arms: Group B: Follistim and Menopur
Drug: Leuprolide — Promotes endogenous LH surge signaling oocyte maturation followed by ovulation. This controls timing for oocyte collection.
  Other Names: Lupron; Leuprolide acetate
Procedure: Transvaginal ultrasound guided needle aspiration of oocytes

SUMMARY:
Disprove the null hypothesis as follows:

Among the investigator's egg bank donors undergoing ovulation induction with recombinant FSH medication per treatment protocol outlined below, use of adjunctive LH activity medication Menopur ™ , will result in the same number of mature oocytes recovered and cryopreserved as from egg donors not treated with Menopur™.

Objectives:

Compare efficacy of recombinant FSH (Follistim ™) with and without adjunct LH activity medication Menopur ™ for our volunteer egg bank donors.

Efficacy defined as:

1. #Days of ovarian stimulation to GnRH agonist trigger.
2. Peak serum estradiol level on day of GnRH agonist trigger.
3. Number of follicles >15 mm average diameter on day of GnRH agonist trigger.
4. Number of mature oocytes recovered and cryopreserved.

Study type: Randomized prospective clinical trial.

Patient selection: Voluntary egg donors who have satisfied all screening criteria for FDA and the Michigan Egg Bank: Age range 18-to 39 years. BMI 18 to 25. Resting antral follicle count of 16 or greater. Cycle day 3 FSH <10 mIU/ml. AMH >2.0 ng/ml.

Study design:

Two groups- Group A- Recombinant FSH Follistim only; Group B- Recombinant FSH Follistim and adjunct Menopur. Both groups will use GnRH agonist trigger 36 hours prior to egg retrieval.

Random number generator with patients assigned basd on odd or even numbers.

Number of subjects: 25 in each group. Total of 50 subjects. This takes into account possible cycle cancellation for poor ovarian response or patient elective withdrawal to result in at least 20 subjects in each group completing the study.

Primary measure of outcome: number of mature oocytes recovered and cryopreserved.

Secondary measures of outcome:

1. #Days of ovarian stimulation to GnRH agonist trigger.
2. Peak serum estradiol level on day of GnRH agonist trigger.
3. Number of follicles >15 mm average diameter on day of GnRH agonist trigger.

DETAILED DESCRIPTION:
Background:

The investigator's Center has been studying human oocyte cryopreservation by vitrification since July 1, 2008 (Western Institutional Board Review -WIRB Pro. Nr: 20081080, WIRB Study Nr.: 1100421). The first phase of the investigator's study was to assess efficacy of oocyte cryopreservation among voluntary egg donors with end points for outcomes including rates of oocyte thaw survival, fertilization, embryo development, implantation, clinical pregnancy, live birth and infant health. The rationale for starting with egg donors was that they represent a population of women most likely to have optimal egg quality and a short turnaround time from vitrification to thaw, IVF and embryo transfer into an appropriate egg recipient patient. If the investigator could establish good outcomes when egg quality is optimal, then there would be good hope to provide reliable egg cryopreservation technology to women in need of fertility preservation when facing treatment of cancer; other illnesses for which treatments harm their eggs; women choosing personal egg banking and for women who wish to avoid excess embryo creation on moral or religious grounds.

The investigator's study observations were that outcomes with use of previously cryopreserved donor eggs was equivalent to fresh donor eggs: 90% of mature oocytes survived the thaw, 76% of thawed oocytes fertilized normally with ICSI, 98% of recipient women had a day 5 embryo transfer with one or two embryos transferred, implantation rate of 42%, 60% or recipient women achieved clinical pregnancy, 58% live birth rate and no birth defects have been observed in over 40 babies delivered through this technology at our Center.

In the beginning of 2012, we opened up the second phase of the investigator's study to include women in need of fertility preservation for the indications mentioned above. No outcomes are yet known due to the expected time deferment from oocyte cryopreservation to use. The favorable outcomes from donor egg bank IVF led to the investigator's establishing the Michigan Egg Bank. On October 22, 2012, the American Society for Reproductive Medicine announced a new practice guideline that oocyte cryopreservation technology should be considered mainstream medical therapy and no long be considered experimental medical care. The investigator's closed the WIRB study November, 26, 2012.

Rationale:

Ovarian stimulation for egg donation should be provided offering the safest and simplest process for our egg donors. Avoiding complications of ovarian hyperstimulation syndrome while assuring recruitment and harvest of good quality oocytes is a main goal in caring for the investigator's volunteer egg donors. Use of FSH medications with GnRH antagonist and GnRH agonist trigger is the protocol of choice for all of the investigator's egg donors. The investigator's egg donors have experienced no complications and rapid recovery. GnRH antagonists have been shown to suppress endogenous ovarian androgen synthesis. In using GnRH antagonist, adjunctive LH or low dose hCG combined with FSH medication has been a mainstream assumption to assure sufficient endogenous ovarian testosterone is present as a substrate for estrogen synthesis and normal folliculogenesis.

In an effort to improve patient compliance by simplifying the use of medications for the investigator's egg donors, the investigator wishes to examine the efficacy of recombinant FSH without additional separate medication of adjunct LH activity in the form Menopur ™.

ELIGIBILITY:
Inclusion Criteria:

* Patient selection: women volunteers in good health wishing to serve as egg donors who have satisfied all screening criteria for FDA and the Michigan Egg Bank: Age range 18-to 28 years. BMI 18 to 25. Resting antral follicle count of 16 or greater. Cycle day 3 FSH <10 mIU/ml. AMH >2.0 ng/ml.

Exclusion Criteria:

* Women who do not meet the inclusion criteria. Cigarette smokers. Fail random drug screening tests.

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-04; Primary Completion 2017-02-12 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
number of mature oocytes recovered and cryopreserved. | 2 weeks
  Immediately after egg harvest, The embyrologist performed microscopic examination of oocytes and is able to determine if the oocyte has completed meiosis 1 with the extrusion of the first polar body and has entered the second stage of meiosis. An oocyte of this developmental stage is considered mature and receptive to a sperm.

SECONDARY OUTCOMES:
1) #Days of ovarian stimulation to GnRH agonist trigger. | 2 weeks
  Day 1 is the first day of menotropin therapy. The total number of days is counted from day 1 until the day of GnRH agonist trigger. This determines the total number of days subject is exposed to menotropin therapy.
2) Peak serum estradiol level on day of GnRH agonist trigger | 2 weeks
  Serum estradiol level is tested in the day of GnRH agonist trigger.
Number of follicles >15 mm average diameter on day of GnRH agonist trigger | 2 weeks
  Transvaginal utlrasound measures average diameter of ovarian follicles. Mature follicles have an average diameter of at least 15 mm or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Mersol-Barg, MD, Principal Investigator — Michigan Reproductive Medicine
Locations (1):
- Michigan Reproductive Medicine, Bloomfield Hills, Michigan, United States